CLINICAL TRIAL: NCT03079310
Title: Thoracic Dorsal Spinal Cord Stimulation for the Treatment of Gait and Balance Impairments in Parkinson Disease
Brief Title: Spinal Cord Stimulation for Gait in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107451
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Parkinson Disease; Atypical Parkinsonism
Keywords: spinal cord stimulation; gait analysis; whole-body kinematics; Parkinson's disease; Neuromodulation; Feature extraction
MeSH Terms: conditions — Parkinson Disease | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord stimulation (Experimental): Boston Scientific SCS system
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — Range of pulse widths (200-500 microseconds) and frequencies (30-130 Hz) will be assessed for each patient
  Other Names: Boston Scientific Precision® System

SUMMARY:
Balance and gait impairment increases the risk of falls and contributes to a reduced quality of life and shorter survival in Parkinson disease (PD) and atypical Parkinsonism patients. In preliminary case studies, electrical epidural spinal cord stimulation (SCS) has been shown to significantly improve gait, postural instability, rigidity, and tremor. Controlled studies for optimizing which stimulation settings produce the best clinical response for mobility and gait, and achieving these results chronically are all significant unmet needs. Using quantitative laboratory and mobile technologies to test a range of stimulation settings, this research study aims to determine which SCS parameters or combination of parameters is best suited to effectively alleviate disabling symptoms experienced by each patient.

ELIGIBILITY:
Inclusion Criteria:

* Consenting male and female participants, aged 18 years to 80 years
* Idiopathic PD with II-IV Hoehn-Yahn stage
* A history of frequent falls, gait and balance dysfunction and postural instability
* ON-freezing
* Ability to perform a gait/walking task (under close supervision),
* PD participants referred by Dr. Jog to the functional neurosurgeon for SCS implantation for treatment of their gait and balance dysfunction and/or for their freezing of gait.
* SCS eligibility has been confirmed by neurologist and neurosurgeon
* Patients who receive SCS for their gait and mobility must participate in this study in order to determine which SCS parameters provide the patient with the best outcome for their PD symptoms.
* able to give informed consent
* Able to attend all clinic visits and assessments
* No dementia or psychiatric abnormalities on neuropsychological testing
* No significant secondary causes (such as cerebrovascular disease, normal pressure hydrocephalus, peripheral neuropathy, severe degenerative lower limb or back disease).

  * we had a few devices to include exploratory trial in atypical PD (MSA, PSP, and CBD confirmed diagnosis from clinic).

Exclusion Criteria:

* History of stroke

  * History of ALS or Myasthenia Gravis
  * Offending medications (Lithium, valproate, steroids, amiodarone, beta-adrenergic agonists (e.g. salbutamol).
  * Persons prescribed zonisamide
  * Women reporting that they are pregnant
  * Persons medically unstable with contraindications to SCS will be excluded
  * Previous brain surgery or cardiac pacemaker
  * Eligibility for deep brain stimulation surgery
  * Moderately severe parkinsonism in the context of unstable pharmacological treatment
  * Dementia as assessed by DSM criteria or severe cognitive disturbances
  * Severe psychiatric symptoms (in particular, hallucinations and depression)
  * Bad general health
  * Lack of compliance at follow-up
  * Severe dyskinesias
  * Significant cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Tailored SCS programming | 3 weeks
  Participants following SCS implantation will undergo 3 programming visits. 9 SCS programs will be tested in a repeated fashion on separate days and at different times of the day (morning vs afternoon). The SCS setting(s) to produce the best motor (gait) response will be used by the participant in-home. SCS device will not be used during this time period.
Changes in spatiotemporal gait measures using objective gait analysis | 12 months
  Spatiotemporal gait parameters known to be affected in parkinsonian syndromes will be analyzed over a 12 month period using gait analysis software. Best SCS setting tailored to each participant's gait symptoms will be assessed at 3-, 6- and 12-months time-points.

SECONDARY OUTCOMES:
Changes in UPDRS-III scores | 12 months
  UPDRS-III assessment will be assessed pre-surgery and post-surgery at 3-, 6- and 12-month time-points while participants are OFF/ON-dopaminergic medication and OFF/ON SCS.
Changes in NFOG-Q scores | 12 months
  NFOG-Q scores will be assessed pre-surgery and post-surgery at 3-, 6- and 12-month time-points.
Changes in PDQ-39 scores | 12 months
  PDQ-39 scores will be assessed pre-surgery and post-surgery at 3-, 6- and 12-month time-points.
Changes in ABC scores | 12 months
  ABC scores will be assessed pre-surgery and post-surgery at 3-, 6- and 12-month time-points.
Changes in QoL scores | 12 months
  QoL scores will be assessed pre-surgery and post-surgery at 3-, 6- and 12-month time-points.
DaTscan imaging | 12-months
  Asymmetry and specific binding ratios (SBRs) of the striatal regions of dopamine transporter from I-123 FP-CIT SPECT images will be quantitatively analyzed from pre-surgery and 12-months of SCS use.
Proprioception testing | 12-months
  KINARM and lower leg KINARM type of robot collects reaction time, speed, force, accuracy and trajectory using a robotic object hitting game to assess cognitive and motor skills to be conducted pre-surgery, and post-SCS at 3-, 6- and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — LHSC
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuentes R, Petersson P, Nicolelis MA. Restoration of locomotive function in Parkinson's disease by spinal cord stimulation: mechanistic approach. Eur J Neurosci. 2010 Oct;32(7):1100-8. doi: 10.1111/j.1460-9568.2010.07417.x. PMID 21039949
- [Background] Santana MB, Halje P, Simplicio H, Richter U, Freire MAM, Petersson P, Fuentes R, Nicolelis MAL. Spinal cord stimulation alleviates motor deficits in a primate model of Parkinson disease. Neuron. 2014 Nov 19;84(4):716-722. doi: 10.1016/j.neuron.2014.08.061. Epub 2014 Oct 30. PMID 25447740
- [Background] Jenkinson N, Nandi D, Muthusamy K, Ray NJ, Gregory R, Stein JF, Aziz TZ. Anatomy, physiology, and pathophysiology of the pedunculopontine nucleus. Mov Disord. 2009 Feb 15;24(3):319-28. doi: 10.1002/mds.22189. PMID 19097193
- [Background] Nagatsua T, Sawadab M. L-dopa therapy for Parkinson's disease: past, present, and future. Parkinsonism Relat Disord. 2009 Jan;15 Suppl 1:S3-8. doi: 10.1016/S1353-8020(09)70004-5. PMID 19131039
- [Background] Liu HG, Zhang K, Yang AC, Zhang JG. Deep brain stimulation of the subthalamic and pedunculopontine nucleus in a patient with Parkinson's disease. J Korean Neurosurg Soc. 2015 Apr;57(4):303-6. doi: 10.3340/jkns.2015.57.4.303. Epub 2015 Apr 24. PMID 25932301
- [Background] Stefani A, Lozano AM, Peppe A, Stanzione P, Galati S, Tropepi D, Pierantozzi M, Brusa L, Scarnati E, Mazzone P. Bilateral deep brain stimulation of the pedunculopontine and subthalamic nuclei in severe Parkinson's disease. Brain. 2007 Jun;130(Pt 6):1596-607. doi: 10.1093/brain/awl346. Epub 2007 Jan 24. PMID 17251240
- [Background] Ferraye MU, Debu B, Fraix V, Goetz L, Ardouin C, Yelnik J, Henry-Lagrange C, Seigneuret E, Piallat B, Krack P, Le Bas JF, Benabid AL, Chabardes S, Pollak P. Effects of pedunculopontine nucleus area stimulation on gait disorders in Parkinson's disease. Brain. 2010 Jan;133(Pt 1):205-14. doi: 10.1093/brain/awp229. Epub 2009 Sep 22. PMID 19773356
- [Background] Giladi N, Horak FB, Hausdorff JM. Classification of gait disturbances: distinguishing between continuous and episodic changes. Mov Disord. 2013 Sep 15;28(11):1469-73. doi: 10.1002/mds.25672. PMID 24132835
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Background] Fenelon G, Goujon C, Gurruchaga JM, Cesaro P, Jarraya B, Palfi S, Lefaucheur JP. Spinal cord stimulation for chronic pain improved motor function in a patient with Parkinson's disease. Parkinsonism Relat Disord. 2012 Feb;18(2):213-4. doi: 10.1016/j.parkreldis.2011.07.015. Epub 2011 Aug 23. No abstract available. PMID 21865071
- [Background] Hassan S, Amer S, Alwaki A, Elborno A. A patient with Parkinson's disease benefits from spinal cord stimulation. J Clin Neurosci. 2013 Aug;20(8):1155-6. doi: 10.1016/j.jocn.2012.08.018. Epub 2013 Feb 26. PMID 23453160
- [Background] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Background] Landi A, Trezza A, Pirillo D, Vimercati A, Antonini A, Sganzerla EP. Spinal cord stimulation for the treatment of sensory symptoms in advanced Parkinson's disease. Neuromodulation. 2013 May-Jun;16(3):276-9. doi: 10.1111/ner.12005. Epub 2012 Dec 10. No abstract available. PMID 23227965
- [Background] Yadav AP, Fuentes R, Zhang H, Vinholo T, Wang CH, Freire MA, Nicolelis MA. Chronic spinal cord electrical stimulation protects against 6-hydroxydopamine lesions. Sci Rep. 2014 Jan 23;4:3839. doi: 10.1038/srep03839. PMID 24452435